CLINICAL TRIAL: NCT04238416
Title: Efficacy of Lactulose Plus Intravenous Branched Chain Amino Acids Versus Lactulose Alone in Patients of Acute on Chronic Liver Failure With Overt Hepatic Encephalopathy: A Prospective Randomized Clinical Trial
Brief Title: Intravenous Branched Chain Amino Acids for Hepatic Encephalopathy in ACLF
Acronym: BCAA-ACLF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-08/2019-1336
Record Dates: First submitted 2019-09-28; First posted 2020-01-23 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure
Keywords: branched chain amino acids; hepatic encephalopathy; lactulose; acute on chronic liver failure; bispectral index
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure | interventions — Amino Acids, Branched-Chain; Lactulose

STUDY DESIGN:
Intervention Model Description: Prospective interventional cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV BCAA + Lactulose (Experimental): IV Branched Chain Amino Acids - 500mL once daily for 3 days plus Lactulose
  Interventions: Drug: Branched chain amino acid; Drug: Lactulose
- Lactulose alone (Active Comparator): Oral Lactulose alone
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Branched chain amino acid — Intravenous branched chain amino acids will be given for 3 days to patients in experimental arm
  Arms: IV BCAA + Lactulose
Drug: Lactulose — Oral lactulose will be given to patients in both arms

SUMMARY:
This study analyses the effect of intravenous branched chain amino acids (BCAA) on overt HE in patients with ACLF. The investigators plan to study the efficacy of combining intravenous BCAA with lactulose versus lactulose alone in the medical management of overt HE in patients with ACLF and its impact on overall survival and improvement in grade of HE.

DETAILED DESCRIPTION:
Acute on chronic liver failure (ACLF) is a distinct clinical entity in the spectrum of chronic liver disease associated with high short term mortality. Hepatic encephalopathy (HE) is commonly seen in patients with ACLF and its treatment mainly involves non-absorbable disaccharides (lactulose/lactitol).Treatment of HE in ACLF is based on extrapolation of data available from cirrhotic patients. No studies have compared different treatment options for HE in patients with ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Either gender
3. Patients with ACLF (CANONIC definition) of any aetiology with HE ≥grade 2 as per West-Haven Criteria or Hepatic encephalopathy scoring algorithm (HESA)

Exclusion Criteria:

1. Those who do not consent to participate in the study
2. Patients with structural brain lesions or stroke
3. Inability to obtain informed consent from patient or relatives
4. Severe preexisting cardiopulmonary disease
5. Renal dysfunction (S. Creatinine ≥ 2mg/dL)
6. Pregnancy/Lactation
7. Post liver transplant patients
8. HIV infection
9. Patients who are on psychoactive drugs, like sedatives or antidepressants
10. Patients who are too sick to carry out the protocol

As the study was carried out during the peak of the COVID-19, patients who developed COVID-19 after randomization were excluded from the analysis as they were shifted to dedicated COVID-19 ICU's.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement of Survival | At day day 28
  All cause Mortality assessment
Improvement of encephalopathy by ≥ 1 grade | 72 hours
  Improvement in hepatic encephalopathy

SECONDARY OUTCOMES:
Reduction in level of ammonia | 48 and 72 hours
Reduction of consciousness recovery time among survivors | 30 days
Prolongation of time to death among non-survivors | 30 days
Prevention/reduction of cerebral edema based on optic nerve sheath diameter | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shawcross DL, Sharifi Y, Canavan JB, Yeoman AD, Abeles RD, Taylor NJ, Auzinger G, Bernal W, Wendon JA. Infection and systemic inflammation, not ammonia, are associated with Grade 3/4 hepatic encephalopathy, but not mortality in cirrhosis. J Hepatol. 2011 Apr;54(4):640-9. doi: 10.1016/j.jhep.2010.07.045. Epub 2010 Dec 1. PMID 21163546
- [Background] Donovan JP, Schafer DF, Shaw BW Jr, Sorrell MF. Cerebral oedema and increased intracranial pressure in chronic liver disease. Lancet. 1998 Mar 7;351(9104):719-21. doi: 10.1016/S0140-6736(97)07373-X. PMID 9504517
- [Background] Albrecht J, Norenberg MD. Glutamine: a Trojan horse in ammonia neurotoxicity. Hepatology. 2006 Oct;44(4):788-94. doi: 10.1002/hep.21357. PMID 17006913
- [Background] Norenberg MD, Martinez-Hernandez A. Fine structural localization of glutamine synthetase in astrocytes of rat brain. Brain Res. 1979 Feb 2;161(2):303-10. doi: 10.1016/0006-8993(79)90071-4. PMID 31966
- [Background] Albrecht J, Dolinska M, Hilgier W, Lipkowski AW, Nowacki J. Modulation of glutamine uptake and phosphate-activated glutaminase activity in rat brain mitochondria by amino acids and their synthetic analogues. Neurochem Int. 2000 Apr;36(4-5):341-7. doi: 10.1016/s0197-0186(99)00142-4. PMID 10733001
- [Background] Laake JH, Takumi Y, Eidet J, Torgner IA, Roberg B, Kvamme E, Ottersen OP. Postembedding immunogold labelling reveals subcellular localization and pathway-specific enrichment of phosphate activated glutaminase in rat cerebellum. Neuroscience. 1999;88(4):1137-51. doi: 10.1016/s0306-4522(98)00298-x. PMID 10336125
- [Background] Cordoba J, Ventura-Cots M, Simon-Talero M, Amoros A, Pavesi M, Vilstrup H, Angeli P, Domenicali M, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of EASL-CLIF Consortium. Characteristics, risk factors, and mortality of cirrhotic patients hospitalized for hepatic encephalopathy with and without acute-on-chronic liver failure (ACLF). J Hepatol. 2014 Feb;60(2):275-81. doi: 10.1016/j.jhep.2013.10.004. Epub 2013 Oct 12. PMID 24128414
- [Result] Fischer JE, Rosen HM, Ebeid AM, James JH, Keane JM, Soeters PB. The effect of normalization of plasma amino acids on hepatic encephalopathy in man. Surgery. 1976 Jul;80(1):77-91. PMID 818729
- [Result] Dam G, Aamann L, Vistrup H, Gluud LL. The role of Branched Chain Amino Acids in the treatment of hepatic Encephalopathy. J Clin Exp Hepatol. 2018 Dec;8(4):448-451. doi: 10.1016/j.jceh.2018.06.004. Epub 2018 Jun 27. PMID 30568347
- [Result] Rossi-Fanelli F, Riggio O, Cangiano C, Cascino A, De Conciliis D, Merli M, Stortoni M, Giunchi G. Branched-chain amino acids vs lactulose in the treatment of hepatic coma: a controlled study. Dig Dis Sci. 1982 Oct;27(10):929-35. doi: 10.1007/BF01316578. PMID 6749458
- [Result] Gluud LL, Dam G, Les I, Cordoba J, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2015 Feb 25;(2):CD001939. doi: 10.1002/14651858.CD001939.pub2. PMID 25715177
- [Derived] Mehtani R, Premkumar M, Garg S, Kajal K, Kulkarni AV, Duseja AK, Dhiman RK, De A, Verma N, Taneja S, Rathi S, Singh V, Chakma J, Soni SL, Kakkar A, Kapila AT, Ahuja CK, Divyaveer S, Praharaj D. Intravenous BCAA Infusion Does Not Lead to a Sustained Recovery From Overt HE in ACLF - An Open Label Randomized Clinical Trial. J Clin Exp Hepatol. 2023 Nov-Dec;13(6):977-988. doi: 10.1016/j.jceh.2023.05.015. Epub 2023 Jun 1. PMID 37975059